CLINICAL TRIAL: NCT00521105
Title: Assessment of an Alternative Model Using Telemedicine Follow-up of Children and Adolescents With Type 1 Diabetes
Brief Title: Assessment of an Alternative Model of Follow-up of Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Dr. Danièle Pacaud, Pediatric Endocrinologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AR-2-05-1823-DP
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Telemedicine; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Participants will be seen every 3-4 months with a physician-only visit alternating with a multidisciplinary visit (MD, RN and RD). This is the current standard of practice.
- 2 (Experimental): Participants will be seen every 3-4 months with a phone contact, with the diabetes nurse educator, alternating with a multidisciplinary visit (MD, RN and RD).
  Interventions: Other: Virtual visit

INTERVENTIONS:
Other: Virtual visit — Participants will alternate between a multidisciplinary visit (MD, RN and RD) and a phone contact with the diabetes nurse educator (the phone contact will replace the physician-only visit). Prior to the phone contact, transmission of information from the participant will be sent through either fax or a web browser.
  Arms: 2

SUMMARY:
The purpose of the study is to look at the effect of replacing the physician only visit by a transmission of information on the participant's current diabetes management and blood glucose monitoring results followed by a phone contact by the diabetes nurse educator. The study will also measure the effect on diabetes control (HbA1c), satisfaction with care, resource utilisation, and costs to the health care system and to the participant.

We hypothesize that replacement of the physician-only visit by a virtual visit will not result in worsening of the medical outcomes and that it will result in a reduction in medical resources utilization and costs for families while increasing the satisfaction with care.

DETAILED DESCRIPTION:
Improved metabolic control reduces both the onset and progression of diabetes-related complications in adults and adolescents with type 1 diabetes. Frequency of contact with the medical care team has been associated with better control. Both the American Diabetes Association and Canadian Diabetes Association recommend regular quarterly visits. However, the increase in case loads and the limited manpower available forces us to look at alternative models of care. A model of care in which medical visits alternate between a face to face multidisciplinary visits and a virtual visit done via fax or e-mail communication and a phone call may be advantageous to both the patient and the medical care team. For the patient and his family, this model would decrease time away from school and work, travel inconveniences and costs. For the medical care team it may decrease time per patient and therefore increase the number of patients served with the same resources.

ELIGIBILITY:
Inclusion Criteria:

* Children: 17 years of age or less
* Diagnosis of Type 1 Diabetes for at least 12 months
* Currently being followed at the Alberta Children's Hospital Diabetes Clinic.

Exclusion Criteria:

* Compromised metabolic control (HbA1c > 10%)
* Uncontrolled hypo or hyperthyroidism
* Uncontrolled celiac disease
* Language or psychosocial barrier preventing the family from completing the study
* Diabetes duration of less than 1 year
* Participation in other clinical trials with specified clinic visits.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Medical outcomes: HbA1c, rates of severe hypoglycemia, rates of DKA | 1 year

SECONDARY OUTCOMES:
Resource utilization: physicians, nurses, and dietitians, emergency room visits | 1 year
Family satisfaction with diabetes care | 1 year
Associated costs to the family (time away from school and work, travel, etc) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danièle Pacaud, MD, Principal Investigator — University of Calgary
Locations (1):
- Endocrine Clinic, Alberta Children's Hospital, Calgary, Alberta, Canada